CLINICAL TRIAL: NCT04766008
Title: Metformin Continuation Safety in Diabetic Patients Undergoing Coronary Angiography
Brief Title: Metformin in Diabetic Patients Undergoing Coronary Angiography
Acronym: NO-STOP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Humanitas Hospital, Italy (Other)
Responsible Party: Principal Investigator, Giulio Stefanini, Professor, Humanitas Hospital, Italy
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20190918
Record Dates: First submitted 2021-01-26; First posted 2021-02-23 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Diabetes Mellitus; Coronary Artery Disease; Lactic Acidosis With Diabetes Mellitus; Contrast-induced Nephropathy; Metformin Associated Lactic Acidosis
Keywords: metformin; coronary angiography; diabetes mellitus; lactic acidosis
MeSH Terms: conditions — Diabetes Mellitus; Coronary Artery Disease; Acidosis, Lactic | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Metformin continuation (Experimental)
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Diabetic patients treated with metformin undergoing coronary angiography will not suspend metformin before and after PCI.

SUMMARY:
The present study aims to evaluate the strict application of the 2018 European Society of Cardiology guidelines on myocardial revascularization, that recommends to check renal function if patients have taken metformin immediately before angiography and withhold metformin if renal function deteriorates.

The aim of this study is to assess the safety of metformin in diabetic patients undergoing coronary angiography in terms of risk of lactic acidosis and to individuate eventual predictors of augmented lactate after coronary angiography.

DETAILED DESCRIPTION:
The study is designed as an open-label (both physician and participant know that metformin will not be discontinued before PCI and in the following 48 hours), prospective, single arm study.

In our historical cohort of diabetic patients taking metformin, we observed a mean value of lactate of 1.2+0.7 mmol/l.

A total of 150 patients will be enrolled. Patients with any deviations from the study protocol will be enrolled in a parallel observational registry.

The study consists of a screening phase, a 30-day observational phase, and an end-of-follow-up visit or phone interview. The total duration of participation in the study for each participant is approximately 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients treated with metformin undergoing coronary angiography.

Exclusion Criteria:

* Known coronary anatomy with planned complex percutaneous coronary intervention with high probability of large amount of contrast use (3.7 * estimated glomerular filtration rate; e.g.: 167 ml in a patients with an eGFR of 45 ml/min/1.73m2).
* Moderate to severe impairment of renal function (eGFR<45 ml/min).
* Moderate to severe impairment of liver function (Child-Pugh class B or C).
* Severely impaired left ventricular ejection fraction (LVEF <35%).
* Patients undergoing primary percutaneous coronary intervention (i.e., patients presenting with ST elevation myocardial infarction).
* Severe to very severe chronic obstructive pulmonary disease (GOLD class 3 to 4).
* Patients scheduled for cardiac surgery in the following 5 days.
* Inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-01-15 (Actual); Primary Completion 2022-04-11 (Actual); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Increase in lactate of 20% | From preprocedural values (same day of the coronary angiography) to 72 hours after coronary angiography
  Lactate will be measured from a venous sampling at three different time points, before coronary angiography, the day after (not mandatory) and 3 days after coronary angiography

SECONDARY OUTCOMES:
Contrast-associated acute kidney injury after coronary angiography. | From 0 to 7 days after coronary angiography
  Contrast-associated acute kidney injury was defined according to the KDIGO definition: increase in serum creatinine of 0.3 mg/dl within 48 hours from coronary angiography or >50% within 7 days (if creatinine after 7 days is available) or urine output of <0.5 ml/kg/hour for at least 6 hours
Metformin associated lactic acidosis | At 24 and 72 hours after coronary angiography
  Lactic acidosis was defined as pH less than or equal to 7.35 and lactatemia greater than 2.2 mmol/L

OTHER OUTCOMES:
Death | Within 30 days after the index coronary angiography
  All cause mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Humanitas Research Hospital, Rozzano, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided
The data that support the findings of this study will be available from the corresponding author on reasonable request.

REFERENCES:
- [Background] Pfisterer ME, Zellweger MJ. Therapies for type 2 diabetes and coronary artery disease. N Engl J Med. 2009 Oct 1;361(14):1407; author reply 1409-10. doi: 10.1056/NEJMc091419. No abstract available. PMID 19797290
- [Background] Bailey CJ, Turner RC. Metformin. N Engl J Med. 1996 Feb 29;334(9):574-9. doi: 10.1056/NEJM199602293340906. No abstract available. PMID 8569826
- [Background] Maznyczka A, Myat A, Gershlick A. Discontinuation of metformin in the setting of coronary angiography: clinical uncertainty amongst physicians reflecting a poor evidence base. EuroIntervention. 2012 Jan;7(9):1103-10. doi: 10.4244/EIJV7I9A175. PMID 21959259
- [Background] Timmer JR, Ottervanger JP, de Boer MJ, Dambrink JH, Hoorntje JC, Gosselink AT, Suryapranata H, Zijlstra F, van 't Hof AW; Zwolle Myocardial Infarction Study Group. Hyperglycemia is an important predictor of impaired coronary flow before reperfusion therapy in ST-segment elevation myocardial infarction. J Am Coll Cardiol. 2005 Apr 5;45(7):999-1002. doi: 10.1016/j.jacc.2004.12.050. PMID 15808754
- [Background] Mehran R, Dangas GD, Weisbord SD. Contrast-Associated Acute Kidney Injury. Reply. N Engl J Med. 2019 Sep 26;381(13):1296-1297. doi: 10.1056/NEJMc1908879. No abstract available. PMID 31553855
- [Background] Neumann FJ, Sousa-Uva M, Ahlsson A, Alfonso F, Banning AP, Benedetto U, Byrne RA, Collet JP, Falk V, Head SJ, Juni P, Kastrati A, Koller A, Kristensen SD, Niebauer J, Richter DJ, Seferovic PM, Sibbing D, Stefanini GG, Windecker S, Yadav R, Zembala MO. 2018 ESC/EACTS Guidelines on myocardial revascularization. EuroIntervention. 2019 Feb 20;14(14):1435-1534. doi: 10.4244/EIJY19M01_01. No abstract available. PMID 30667361
- [Background] Parra D, Legreid AM, Beckey NP, Reyes S. Metformin monitoring and change in serum creatinine levels in patients undergoing radiologic procedures involving administration of intravenous contrast media. Pharmacotherapy. 2004 Aug;24(8):987-93. doi: 10.1592/phco.24.11.987.36131. PMID 15338847
- [Background] Nawaz S, Cleveland T, Gaines PA, Chan P. Clinical risk associated with contrast angiography in metformin treated patients: a clinical review. Clin Radiol. 1998 May;53(5):342-4. doi: 10.1016/s0009-9260(98)80005-6. PMID 9630271
- [Background] Laskey WK, Jenkins C, Selzer F, Marroquin OC, Wilensky RL, Glaser R, Cohen HA, Holmes DR Jr; NHLBI Dynamic Registry Investigators. Volume-to-creatinine clearance ratio: a pharmacokinetically based risk factor for prediction of early creatinine increase after percutaneous coronary intervention. J Am Coll Cardiol. 2007 Aug 14;50(7):584-90. doi: 10.1016/j.jacc.2007.03.058. Epub 2007 Jul 30. PMID 17692741
- [Derived] Chiarito M, Sanz-Sanchez J, Piccolo R, Condello F, Liccardo G, Maurina M, Avvedimento M, Regazzoli D, Pagnotta P, Garcia-Garcia HM, Mehran R, Federici M, Condorelli G, Diez Gil JL, Reimers B, Ferrante G, Stefanini G. Safety of metformin continuation in diabetic patients undergoing invasive coronary angiography: the NO-STOP single arm trial. Cardiovasc Diabetol. 2023 Feb 6;22(1):28. doi: 10.1186/s12933-023-01744-4. PMID 36747244

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-22): https://cdn.clinicaltrials.gov/large-docs/08/NCT04766008/Prot_SAP_000.pdf
  • Informed Consent Form (2019-10-22): https://cdn.clinicaltrials.gov/large-docs/08/NCT04766008/ICF_001.pdf